CLINICAL TRIAL: NCT01731821
Title: A Prospective Randomized Clinical Trial of Two Surgical Techniques for Pancreaticojejunostomy in Patients Undergoing Pancreaticoduodenectomy: Nonstented Stump-closed vs Duct-to-Mucosa Pancreaticojejunostomy
Brief Title: Nonstented Stump-closed vs Duct-to-Mucosa Pancreaticojejunostomy After Pancreaticoduodenectomy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Xian-Jun Yu, Professor and Chair,Department of Pancreatic & Hepatobiliary Surgery, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PCI001
Record Dates: First submitted 2012-11-10; First posted 2012-11-22 (Estimated); Last update posted 2014-12-04 (Estimated); Status verified 2014-12

CONDITIONS: Pancreatic Neoplasms; Biliary Tract Neoplasms; Pancreatitis, Chronic; Duodenal Neoplasms
Keywords: Pancreaticoduodenectomy; Pancreaticojejunostomy
MeSH Terms: conditions — Pancreatic Neoplasms; Biliary Tract Neoplasms; Pancreatitis, Chronic; Duodenal Neoplasms | interventions — Pancreaticojejunostomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nonstented stump-closed anastomosis (Experimental): Nonstented stump-closed anastomosis is used for pancreaticojejunostomy after pancreaticoduodenectomy.
  Interventions: Procedure: pancreaticojejunostomy
- Duct-to-mucosa anastomosis (Active Comparator): Duct-to-mucosa technique is used for pancreaticojejunostomy after pancreaticoduodenectomy.
  Interventions: Procedure: pancreaticojejunostomy

INTERVENTIONS:
Procedure: pancreaticojejunostomy — Nonstented stump closed pancreaticojejunostomy:
  Close the pancreatic stump with interrupted inverting sutures around the "papillary-like" pancreatic duct.
  A small full-thickness enterotomy was penetrated on the jejunal wall for connecting to the "papillary-like" pancreatic duct by placing 4-6 sutures from the "periductal" parenchyma to the whole-layer jejunum hole. After that, interrupted sutures between the front wall of pancreatic stump and the seromuscular jejunum were performed by 4-0 absorbable sutures to complete the anastomosis.
  Duct-to-mucosa pancreaticojejunostomy:Two layer anatomosis with "Duct-to-Mucosa" pancreaticojejunostomy is performed by suturing the pancreatic parenchyma to the jejunal seromuscular layer and no stenting tube was used.

SUMMARY:
Pancreaticojejunostomy is the key procedure of pancreaticoduodenectomy. The aim of our study is to investigate a new pancreaticojejunal (PJ) anastomosis procedure named "nonstented stump-closed pancreaticojejunostomy" in pancreatoduodenectomy, which could provide a feasible option to pancreatic surgeons for patients with pancreaticoduodenectomy.

DETAILED DESCRIPTION:
Pancreaticoduodenectomy is a standard surgical approach for resectable pancreatic tumors and periampullary tumors. It is considered a safe procedure resulting from the continuous improvement in surgical techniques over the years. Although postoperative mortality has obviously decreased, pancreatic fistula is still a major challenge in pancreatic surgery and remains the major cause of postoperative morbidity and mortality after pancreaticoduodenectomy(PD), ranging from 5% to 30%.

Many risks factors have been shown to cause pancreatic fistula(PF) after the operation, including advanced age, prolonged operation time, intraoperative hemorrhage, BMI, soft pancreas, size of the main pancreatic duct and texture of the remnant pancreas. Among them, soft pancreatic texture without a dilated main pancreatic duct is regarded as the most important risk factor in predicting pancreatic fistula.

The serious consequences of pancreatic fistula result from the pancreatic juice becoming activated by the bile and intestinal fluid, which will eventually corrupt the PJ anastomosis and the surrounding normal tissues. The corrosion of the vasculature will lead to lethal hemorrhage, which is the main cause of mortality after pancreaticoduodenectomy. Furthermore, pancreatin, together with the bacteria in the alimentary tract, will lead to intra-abdominal infection and abscess. To reduce the pancreatic fistula rate, several techniques have been described as alternatives to the conventional PJ anastomosis. Duct-to-mucosa sutures, binding pancreaticojejunostomy and end-to-side invaginated fashion are widely used in the current clinical setting. Some non-randomized studies showed that the duct-to-mucosa method was a relatively safe approach. However, the prospective clinical study found that in comparison with the conventional end-to-side anastomosis, duct-to-mucosa did not obviously decrease the incidence of pancreatic fistula as well as other operative complications. The Peng's binding anastomosis technique might be relatively simple to operate and have shorter operative time, but as the raw pancreatic surface is exposed to the jejunal lumen directly after the reconstruction, the activated pancreatic juice might lead to hemorrhage through vascular corrosion. Moreover, a wide or large pancreatic stump will not fit the size of the jejunal lumen, which could lead to anastomosis ischemia and leakage. The duct-to-mucosa method is not affected by the size of pancreatic remnant and the jejunal lumen. The seromuscular layer of the jejunum covers the pancreatic stump completely and will lower the incidence of postoperative hemorrhage. It was proved to be superior to invagination anastomosis in terms of anastomotic patency and function. Unfortunately, in the cases of small main pancreatic duct or normal soft pancreas, the duct-to-mucosa approach is difficult to operate and takes more surgery time, while simultaneously increasing the incidence of postoperative pancreatic fistula(POPF). Therefore, it is difficult to find a single superior strategy that applies to every case. Selecting an optimal pancreaticojejunal anastomotic method should be based on the different textures of pancreas and the various sizes of the main pancreatic duct.

The postoperative pancreatic fistula (POPF), which determines postoperative mortality, length of hospital stay， is dependent of its definition, and is reported in up to 16% of patients. The purpose of this study is to determine whether the new anastomosis called "nonstented stump-closed" pancreaticojejunostomy can reduce the POPF rate and downgrade compared with the common accepted duct-to-mucosa pancreaticojejunostomy after pancreaticoduodenectomy. This single-centre, open, randomized controlled trail is conducted following International Study Group on Pancreatic Fistula (ISGPF) criteria for pancreatic fistula (PF). The primary endpoint is the POPF rate, and others include overall postoperative complication rate and their severity reoperation rate and hospital stay.

Objectives:

Through the comparison with classic pancreatic duct-to-mucosa anastomosis, to evaluate whether "nonstented stump closed" pancreaticojejunal anastomosis can reduce the pancreatic fistula and other complications incidence; to evaluated the safety and maneuverability.

Patients and methods :all patients diagnosed with periampullar occupations which should be resected through pancreaticoduodenectomy will be evaluated before surgery, including CT,Magnetic Resonance(MR), Ultrasound B ,blood biochemical checks and cardiac and thoracical evaluations. Before the surgery, the patients are divided into two groups by randomization. After the pancreaticoduodenectomy, the randomization number decided the procedure of the pancreaticojejunostomy.

Staging investigations will be standard and will include:

pancreatic enhanced CT; magnetic resonance cholangiopancreatography(MRCP); PET-CT if necessary;

Randomization:

Block randomization will be done using a computer generated sheet. Randomization will be performed 1 day before the operation.

All surgeries will be performed under general anesthesia with epidural analgesia. The surgery will be either performed by or under the direct supervision of pancreatic surgeons with experience in pancreaticojejunostomy surgery. Operative time, blood loss, blood product replacement and all intraoperative details will be recorded in the proforma. Patients will be shifted postoperatively to the anesthesia care unit (PCU) for observation and subsequently to the recovery or high dependency ward once stabilized. Postoperative details including period of postoperative pancreatic fistula,biliary leakage,postoperative haemorrhage,postoperative pancreatitis , hospital stay and other complications will be recorded. Postoperative mortality will be defined as 30-day mortality plus death before discharge after surgery.

Data management: All collected data will be entered into a statistical software package for subsequent analysis

Main research variables:

Primary Outcome :

The primary endpoint will be the postoperative pancreatic fistula(POPF) rate.

Secondary Outcome Measures:

postoperative hospital stay time; anastomosis time; reoperation rate; morbidity

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* 18-80 years old;
* Eastern Cooperative Oncology Group(ECOG) 0-2
* Patients must have undergone pancreaticoduodenectomy.
* Preoperative enhanced CT scan shows respectable or borderline resectable neoplasm
* Without distal metastasis

Exclusion Criteria:

* Patients who have had previous pancreatic body tail resection rese
* immunodeficiency, people infected with HIV
* patients with severe cardiopulmonary function, liver and renal function
* infection without control or active infections
* Pregnant patients.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 308 (Actual)
Dates: Start 2012-10; Primary Completion 2014-06 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
the postoperative pancreatic fistula(POPF) rate | 30 days

SECONDARY OUTCOMES:
postoperative hospital stay time; | 90 days
anastomosis time; | 1 hour
reoperation rate; | 30 days
morbidity and mortality | 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Xian-Jun Yu, M.D., Principal Investigator — Department of Pancreatic & Hepatobiliary Surgery
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Xu J, Zhang B, Shi S, Qin Y, Ji S, Xu W, Liu J, Liu L, Liu C, Long J, Ni Q, Yu X. Papillary-like main pancreatic duct invaginated pancreaticojejunostomy versus duct-to-mucosa pancreaticojejunostomy after pancreaticoduodenectomy: A prospective randomized trial. Surgery. 2015 Nov;158(5):1211-8. doi: 10.1016/j.surg.2015.04.020. Epub 2015 May 30. PMID 26036878